CLINICAL TRIAL: NCT04911634
Title: Laparoscopic Ultrasound Guided Minimal Invasive Excision of Intra-/Retroperitoneal Tumors in Patients Scheduled for Laparotomy: A Pilot Study
Brief Title: Laparoscopic Ultrasound Guided Minimal Invasive Excision of Intra-/Retroperitoneal Tumors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Michael Bau Mortensen, Professor, MD, PhD, DMSc, Odense University Hospital
Other Study IDs: MBM-41
Record Dates: First submitted 2021-05-28; First posted 2021-06-03 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2020-05

CONDITIONS: Laparoscopic Ultrasound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Patients included in the study went through standard preoperative preparation and were informed about potential conversion to open surgery. The procedure started with LUS performed according to the department's standard guidelines (one twelve mm trocar in the midline and one 12 mm trocar in the left upper quadrant) followed by a stepwise scanning of relevant structures (e.g. liver, pancreas, retroperitoneum) with dedicated laparoscopic ultrasound equipment (BK Medical, Herlev, Denmark). If the suspected lesion(s) was detected by LUS in the relevant area (according to preoperative imaging), laparoscopic resection was attempted, and if successful the specimen was removed in an eEndo-bBag (Kebomed, Denmark) through one of the trocars. A second LUS was performed to ensure that no tumor was left behind ("loss-of-lesion(s)").

If any problem occurred during the laparoscopic procedure, the operation was converted to an open procedure. Prophylactic antibiotics were not given routinely but were administered during surgery at the surgeons' discretion.

The intra- and postoperative course and final clinical outcome including pathology reports were retrieved from the patient's electronical records. This included a postoperative follow up of at least 12 months to investigate potential incomplete resection. Postoperative complications were graded according to Dindo-Clavien (17). The pathology reports were retrieved from the Danish Pathology Registry.

ELIGIBILITY:
Inclusion Criteria:

Patients with intra- and retroperitoneal tumor(s) (IRT) detected by imaging (US/CTMR/PET or EUS) and a clinical indication for explorative laparotomy

Exclusion Criteria:

Patients with contraindications for laparoscopy, such as severe adherences were excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients were discussed at the Upper or Lower GI Multidisciplinary Team conferences MDT in order to make sure that only patients where explorative laparotomy was considered the next and only possible clinical step, were referred for the minimal invasive procedure.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2005-01-01 (Actual); Primary Completion 2021-05-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Tumor localization | 12 months
  Positive LUS localization of the tumor(s) in minimum 15 patients
LUS guided resection | 12 months
  A complete LUS guided resection in minimum 15 patients

SECONDARY OUTCOMES:
Complications | 12 months
  No clinical important complications (Dindo-Clavien ≥3) in any of the patients where LUS guided resection was performed and completed
Final diagnosis | 12 months
  A pathological diagnosis was obtained based on the resected tumor(s) in all cases. The LUS guided procedure should obviate the need for (subsequent) open surgery in all patients

CONTACTS AND LOCATIONS:
Locations (1):
- Odense University Hospital, Odense C, Denmark

IPD SHARING:
Plan to Share IPD: No